CLINICAL TRIAL: NCT01367444
Title: A Phase I/IIA Dose Escalation Safety Study of Subretinally Injected SAR422459, Administered to Patients With Stargardt's Macular Degeneration
Brief Title: Phase I/IIA Study of SAR422459 in Participants With Stargardt's Macular Degeneration
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study stopped not for safety reasons. Due to review of clinical development plans and priorities, Sponsor decided to stop development of the product.
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TDU13583; SG1/001/10
Record Dates: First submitted 2011-06-03; First posted 2011-06-07 (Estimated); Results first posted 2020-06-05 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-03

CONDITIONS: Stargardt's Disease
Keywords: Stargardt's Disease
MeSH Terms: conditions — Stargardt Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- SAR422459 (Dose 1) (Experimental): Starting dose of SAR422459 given through subretinal injection
  Interventions: Drug: SAR422459
- SAR422459 (Dose 2) (Experimental): Escalating dose of SAR422459 given through subretinal injection
  Interventions: Drug: SAR422459
- SAR422459 (Dose 3) (Experimental): Maximum tolerated dose (MTD) of SAR422459 given through subretinal injection
  Interventions: Drug: SAR422459

INTERVENTIONS:
Drug: SAR422459 — Pharmaceutical form: sterile solution, 100 microliters (μL) aliquots in 0.3 milliliter (mL) type I borosilicate glass 'V' vials with a butyl stopper and aluminum crimp seal.
  Route of administration: subretinal injection

SUMMARY:
Primary Objective:

To assess the safety and tolerability of ascending doses of SAR422459 in participants with Stargardt's Macular Degeneration (SMD).

Secondary Objective:

To evaluate for possible biological activity of SAR422459.

DETAILED DESCRIPTION:
The total duration per participant was up to 52 weeks, which included 4 week screening period and 48 weeks study period.

At the end of the study, the participants were invited to enter in an open-label safety study (LTS13588-NCT01736592) for long-term follow-up visits including ophthalmological examinations and recording of adverse events (AEs) for up to 15 years.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated written informed consent obtained from the participant and/or the participant's legally acceptable representative.
* Diagnosis of SMD, with at least one pathogenic mutant ABCA4 allele on each chromosome.
* Women of childbearing potential must had a negative pregnancy test at Day -1, and agree to use an effective form of contraception for at least three months, or be surgically sterile or postmenopausal, with the last menstrual period being over two years prior to enrollment.
* Males must agree with their partner to use two forms of contraception for at least three months following SAR422459 administration.
* Participants must agree to not donate blood, organs, tissues or cells for at least three months following SAR422459 administration.
* Participants enrolled in France must be affiliated to or benefit from a social security regimen.

Specific Inclusion Criteria Participant Group A:

* Participants (18 years or older) with advanced SMD.
* Visual acuity less than or equal to (<=) 20/200 in the worst eye.
* Severe cone-rod dysfunction with no detectable or severely abnormal full-field electroretinogram responses.

Specific Inclusion Criteria Participant Group B:

* Participants (18 years or older) with SMD.
* Visual Acuity <=20/200 in the worst eye.
* Abnormal full-field electroretinogram responses.

Specific Inclusion Criteria Participant Group C:

* Participants (18 years or older) with SMD.
* Visual acuity <=20/100 in the worst eye.
* Abnormal full-field electroretinogram responses.

Specific Inclusion Criteria Participant Group D:

* Symptomatic participants (from 6 years to 26 years old) with early or childhood-onset SMD (age at disease onset [less than] <18 years) with at least one pathogenic mutant ABCA4 allele on each chromosome confirmed by direct sequencing and co-segregation analysis within the participant's family.
* Visual acuity of greater than or equal to (>=) 20/200 in both eyes at the time of the screening visit.
* Participants were anticipated to experience rapid deterioration in visual function and/or retinal structure as determined by an annual progression rate in at least one of the following parameters occurring in at least one eye (assessments recorded up to 2 years prior to the screening visit date might be considered to document evidence of rapid deterioration):

  * Loss of >=1 line of Snellen visual acuity (equivalent to 5 early treatment diabetic retinopathy study [ETDRS] letters).
  * Reduction in macular mean sensitivity of >=1.2 decibels (dB) as assessed by microperimetry.
  * Reduction in macular mean sensitivity of >=5 dB or reduction in hill of vision by greater than (>)14 dB-sr as assessed by static perimetry.
  * Enlargement in the area of macular retinal pigment epithelial (RPE) atrophy by fundus autofluorescence at a rate of >=0.5 millimeter square(mm^2).
  * Enlargement in the area of central macular retinal thinning/photoreceptor loss by ocular coherence tomography at a rate of >=0.5 mm^2.
* All eligible participants must demonstrate an ability to understand, willingness to cooperate and ability to reliably perform required study procedures as judged and confirmed by the study investigator.

Specific inclusion criteria Participant Group E:

* Symptomatic participants (between 6 years and 17 years old) with early or childhood-onset SMD with at least one pathogenic mutant ABCA4 allele on each chromosome confirmed by direct sequencing and co-segregation analysis within the participant's family.
* Visual acuity of >=20/100 in both eyes at the time of screening visit.
* Participants were anticipated to experience rapid deterioration in visual function and/or retinal structure as determined by an annual progression rate in at least one of the following parameters occurring in at least one eye (assessments recorded up to 2 years prior to the screening visit date were considered to document evidence of rapid deterioration):

  * Loss of >=1 line of Snellen visual acuity (equivalent to 5 ETDRS letters).
  * Reduction in macular mean sensitivity of >=1.2 dB as assessed by microperimetry.
  * Reduction in macular mean sensitivity of >=5 dB or reduction in hill of vision by >14 dB-sr as assessed by static perimetry.
  * Enlargement in the area of macular RPE atrophy by fundus autofluorescence at a rate of >=0.5 mm^2.
  * Enlargement in the area of central macular retinal thinning/photoreceptor loss by ocular coherence tomography at a rate of >=0.5 mm^2.
* All eligible participants demonstrated an ability to understand, willingness to cooperate and ability to reliably perform required study procedures as judged and confirmed by the study investigator.

Exclusion Criteria:

* Pre-existing eye conditions that would preclude the planned surgery or interfere with the interpretation of study outcome measures.
* Cataract surgery with intraocular lens implantation within 6 months of enrolment.
* Aphakia or prior vitrectomy in the study eye.
* Concomitant systemic diseases including those in which the disease itself, or the treatment for the disease, can alter ocular function.
* Any intraocular surgery or laser in either eye planned within 6 months of Day 0.
* Any contraindication to pupil dilation in either eye.
* Any known allergy to any component of the delivery vehicle or diagnostic agents used during the study, or medications planned for use in the perioperative period particularly topical, injected or systemic corticosteroids.
* Any injectable intravitreal treatment to the treated eye or intravitreal device in the treated eye within 6 months prior to screening.
* Any periocular injections of corticosteroids to the treated eye within 4 months prior to screening.
* Laboratory test abnormalities or abnormalities in electrocardiogram, chest X-rays that in the opinion of the Principal Investigator would make the participant unsuitable for participation in the study.
* Significant intercurrent illness or infection during the 28 days prior to enrolment.
* Pre-menopausal or non-surgically sterile women who were unwilling to use an effective form of contraception such as the contraceptive pill or intrauterine device.
* Alcohol or other substance abuse.
* Contraindications to use of anesthesia (local or general, as appropriate).
* Concurrent anti-retroviral therapy that would inactivate the investigational agent.
* History of any investigational agent within 28 days prior to SAR422459 administration.
* Participation in a prior ocular gene transfer therapy study.
* Enrolment in any other clinical treatment study throughout the duration of the SAR422459 study.
* Current or anticipated treatment with anticoagulant therapy or the use of anticoagulation therapy within the four weeks prior to surgery.
* A past medical history of human immunodeficiency virus or hepatitis A, B, or C infection.
* Women who were pregnant or were breastfeeding.
* History or signs consistent with unilateral amblyopia (strabismic, anisometropic, or stimulus deprivation).

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2011-06-08 (Actual); Primary Completion 2019-08-16 (Actual); Study Completion 2019-08-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Yang, MD, Principal Investigator — Oregon Health & Science University, Portland, Oregon; Jose-Alain Sahel, MD. Ph.D, Principal Investigator — Hopital Nationale des Quinze-Vingt, Paris France
Locations (5):
- United States (4):
  - Investigational Site Number 840002, Miami, Florida
  - Investigational Site Number 840005, Iowa City, Iowa
  - Investigational Site Number 840001, Portland, Oregon
  - Investigational Site Number 840004, Houston, Texas
- Investigational Site Number 250001, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Davis JL. The Blunt End: Surgical Challenges of Gene Therapy for Inherited Retinal Diseases. Am J Ophthalmol. 2018 Dec;196:xxv-xxix. doi: 10.1016/j.ajo.2018.08.038. Epub 2018 Sep 5. PMID 30194931
- [Derived] Parker MA, Choi D, Erker LR, Pennesi ME, Yang P, Chegarnov EN, Steinkamp PN, Schlechter CL, Dhaenens CM, Mohand-Said S, Audo I, Sahel J, Weleber RG, Wilson DJ. Test-Retest Variability of Functional and Structural Parameters in Patients with Stargardt Disease Participating in the SAR422459 Gene Therapy Trial. Transl Vis Sci Technol. 2016 Oct 1;5(5):10. doi: 10.1167/tvst.5.5.10. eCollection 2016 Oct. PMID 27730010

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The Study was conducted in France and the United States. The trial was ended prematurely and the end of trial date declaration to health authorities was 16-August-2019.
Pre-assignment Details: A total of 35 participants who had Stargardt's Macular Degeneration (SMD) were screened, out of which 27 participants were enrolled in 7 cohorts (Cohorts 1 to 7).
Groups:
- Cohort 1: Participants (aged greater than or equal to [>=] 18 years) with advanced SMD, and visual acuity (VA) less than or equal to (<=) 20/200 in the worst eye and severe cone-rod dysfunction with no detectable or severely abnormal full-field electroretinography (ERG) responses, received SAR422459 at lowest target dose level 1.8*10^5 transducing units (TU)/study eye.
- Cohort 2: Participants (aged >=18 years) with SMD, and VA <=20/200 in the worst eye with abnormal full-field ERG responses, received SAR422459 at lowest target dose level 1.8*10^5 TU/study eye.
- Cohort 3: Participants (aged >=18 years) with SMD, and VA <=20/200 in the worst eye with abnormal full-field ERG responses, received SAR422459 at escalated target dose level 6*10^5 TU/study eye.
- Cohort 4: Participants (aged >=18 years) with SMD, and VA <=20/200 in the worst eye with abnormal full-field ERG responses, received SAR422459 at target dose level 1.8*10^6 TU/study eye.
- Cohort 5: Participants (aged >=18 years) with SMD, and VA <=20/100 in the worst eye with abnormal full-field ERG responses, received SAR422459 at highest target dose level 1.8*10^6 TU/study eye.
- Cohort 6: Participants (aged 6 to 26 years) with symptomatic early or childhood-onset SMD, and VA >=20/200 in both eyes at the time of the screening visit and anticipated to experience rapid deterioration in visual function and/or retinal structure, received SAR422459 at highest target dose level 1.8*10^6 TU/study eye.
- Cohort 7: Pediatric participants (aged 6 to 17 years) with symptomatic SMD, and VA >=20/100 in both eyes at the time of the screening visit and anticipated to experience rapid deterioration in visual function and/or retinal structure, received SAR422459 at highest target dose level 1.8*10^6 TU/study eye.
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6 | Cohort 7
Started | 4 | 4 | 4 | 4 | 6 | 4 | 1
Completed | 4 | 4 | 4 | 4 | 6 | 4 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Cohort 1: Participants (aged >=18 years) with advanced SMD, and VA <=20/200 in the worst eye and severe cone-rod dysfunction with no detectable or severely abnormal full-field ERG responses, received SAR422459 at lowest target dose level 1.8*10^5 TU/study eye.
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6 | Cohort 7 | Total
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 6 | 4 | 1 | 27
Age, Continuous [Median (Full Range); unit: years] | 55.5 [32 to 66] | 40 [30 to 63] | 44.5 [35 to 60] | 40 [28 to 56] | 28 [24 to 41] | 23 [21 to 37] | 16 [16 to 16] | 36 [16 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4 | 0 | 2 | 2 | 1 | 13
  Male | 3 | 1 | 0 | 4 | 4 | 2 | 0 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  White | 4 | 4 | 3 | 3 | 6 | 4 | 1 | 25
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any unfavorable and unintended physical sign, symptom, or laboratory parameter that developed or worsened in severity during the course of the study, whether or not considered related to the investigational product. The TEAEs were defined as any event that started or increased in severity after the participant received investigational medicinal product (IMP), including abnormal laboratory results, electrocardiogram, etc.
Time Frame: From Baseline to Week 48
Population: Analysis was performed on all participants with SMD who were included in the study.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6 | Cohort 7
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 6 | 4 | 1
percentage of participants | 100 | 100 | 100 | 100 | 100 | 100 | 100

2. Primary Outcome: Percentage of Participants With TEAEs by Severity
Description: An AE was any unfavorable and unintended physical sign, symptom, or laboratory parameter that developed or worsened in severity during the course of the study, whether or not considered related to the investigational product. For each AE, the severity was categorized as either mild, moderate or severe where 'mild' was defined as discomfort noticed but did not interfere with the participant's daily routines (an annoyance), 'moderate' was defined as some impairment of function, not hazardous to health (uncomfortable or embarrassing), and 'severe' was defined as significant impairment of function, hazardous to health (incapacitating).
Time Frame: From Baseline to Week 48
Population: Analysis was performed on all participants with SMD who were included in the study.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6 | Cohort 7
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 6 | 4 | 1
percentage of participants
  Mild | 100 | 100 | 100 | 100 | 100 | 100 | 100
  Moderate | 0 | 50 | 25 | 25 | 33 | 75 | 100
  Severe | 0 | 0 | 0 | 25 | 17 | 25 | 0

ADVERSE EVENTS:
Time Frame: All AEs were collected from time of first dose of study drug up to end of study (Week 48) regardless of seriousness or relationship (causality) to IMP.
Description: Reported AEs were TEAEs that developed/worsened during the 'on treatment period' (from Day 0 to Week 48). Analysis was performed on all participants with SMD who were included in the study.
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6 | Cohort 7
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4 | 0/4 | 0/4 | 0/6 | 0/4 | 0/1
Serious Adverse Events (participants affected / at risk) | 1/4 | 0/4 | 0/4 | 0/4 | 0/6 | 1/4 | 1/1
Other Adverse Events (participants affected / at risk) | 4/4 | 4/4 | 4/4 | 4/4 | 6/6 | 4/4 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=4) | Cohort 2 (N=4) | Cohort 3 (N=4) | Cohort 4 (N=4) | Cohort 5 (N=6) | Cohort 6 (N=4) | Cohort 7 (N=1)
Chorioretinopathy (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Uveitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Intraocular pressure increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=4) | Cohort 2 (N=4) | Cohort 3 (N=4) | Cohort 4 (N=4) | Cohort 5 (N=6) | Cohort 6 (N=4) | Cohort 7 (N=1)
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ventricular extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Anterior chamber cell (Eye disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Anterior chamber inflammation (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cataract (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Chalazion (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Choroidal effusion (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Conjunctival haemorrhage (Eye disorders) | 3 | 2 | 2 | 1 | 3 | 0 | 0
Corneal disorder (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Diplopia (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dyschromatopsia (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Eye discharge (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Eye disorder (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eye inflammation (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Eye irritation (Eye disorders) | 0 | 0 | 0 | 1 | 2 | 0 | 0
Eye pain (Eye disorders) | 2 | 2 | 1 | 0 | 1 | 0 | 1
Eye pruritus (Eye disorders) | 0 | 1 | 2 | 0 | 2 | 0 | 0
Eyelid irritation (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypotony of eye (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Keratic precipitates (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Macular fibrosis (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Macular oedema (Eye disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Necrotising retinitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ocular hyperaemia (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ocular hypertension (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Photopsia (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Retinal disorder (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Retinal haemorrhage (Eye disorders) | 0 | 1 | 0 | 1 | 1 | 2 | 0
Retinal tear (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Serous retinal detachment (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Subretinal fibrosis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Subretinal fluid (Eye disorders) | 1 | 1 | 1 | 0 | 2 | 0 | 0
Trichiasis (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Uveitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Visual impairment (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Vitreous detachment (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vitreous floaters (Eye disorders) | 1 | 0 | 1 | 0 | 2 | 0 | 0
Vitreous haemorrhage (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Xanthopsia (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dental caries (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Asthenia (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Conjunctivitis (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Conjunctivitis viral (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea infectious (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ear infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 2 | 2 | 1 | 0 | 1 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Cartilage injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Corneal abrasion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tongue injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Colour vision tests abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fundoscopy abnormal (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Intraocular pressure decreased (Investigations) | 0 | 1 | 0 | 1 | 2 | 0 | 0
Intraocular pressure increased (Investigations) | 2 | 3 | 2 | 1 | 0 | 0 | 1
Monoclonal immunoglobulin present (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Visual field tests abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 1 | 1 | 0 | 1 | 1 | 2 | 1
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Visual field defect (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Glycosuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Leukocyturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
The planned analysis was adjusted and carried out on the available safety data collected before the Sponsor's decision to stop SAR422459 development prematurely.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2018-11-29): https://cdn.clinicaltrials.gov/large-docs/44/NCT01367444/Prot_000.pdf
  • Statistical Analysis Plan (2019-09-16): https://cdn.clinicaltrials.gov/large-docs/44/NCT01367444/SAP_001.pdf